CLINICAL TRIAL: NCT04062500
Title: Registry for Longitudinal Mortality and Therapy in Patients With Heart Failure (GREARTWAL Study)
Brief Title: Registry for Longitudinal Mortality and Therapy in Patients With Heart Failure
Acronym: GREARTWAL
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Beijing Chao Yang Hospital (Other); First Hospital of China Medical University (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other); Xuhui Central Hospital, Shanghai (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Shaanxi University of Chinese Medicine (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, MD, pHD, Director of Cardiovascular Department, Shanghai 10th People's Hospital
Other Study IDs: GREARTWAL
Record Dates: First submitted 2019-08-09; First posted 2019-08-20 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Heart Failure,prognostic, registry
MeSH Terms: conditions — Heart Failure | interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human serum from enrolled patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with heart failure: patients treated in the hospital for acute heart failure in China
  Interventions: Other: Mortality and Rehospitalization rate

INTERVENTIONS:
Other: Mortality and Rehospitalization rate — Mortality and Re-hospitalization of acute decompensated heart failure

SUMMARY:
The purpose of this registry is to compile a large clinical database on the medical management of patients hospitalized with acute heart failure, using information collected from hospitals across China.

DETAILED DESCRIPTION:
Registry for Longitudinal mortality and therapy in patients with Heart Failure is a large, multicenter, prospective, open-label registry of the management of patients treated in the hospital for acute heart failure in China. The objective of this study is to investigate the clinical features and prognosis of patients with heart failure, and discover the characteristics of high-risk heart failure patients, and elucidate critical factors which predict the development and outcomes of symptomatic heart failure patients.

1. To elucidate the clinical characteristics and prognostic risks of patients with heart failure.
2. To study the characteristics of high-risk heart failure patients and predict the key factors for the development of symptomatic heart failure patients.
3. To elucidate the compliance of patients with heart failure and the incidence of adverse drug effects.
4. To investigate the effect of self-management on outcomes in patients with heart failure.
5. To elucidate critical factors associated with the development and outcomes of heart failure.
6. To investigate hospitalization expenses for heart failure.

ELIGIBILITY:
Inclusion Criteria:

- 1. 18 years and older. 2. Meet the diagnostic criteria of China 2018 or JACC/AHA 2017 or ESC 2016 heart failure guidelines.

3. Agree to be tested and sign an informed consent certificate.

Exclusion Criteria:

* 1. Age<18 years old. 2. Patients who refused to participate. 3. Patients may have a life expectancy of less than 1 years due to non- heart failure clinical conditions.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality of acute decompensated heart failure | 10 years
  In-hospital and Annual mortality
Re-hospitalization rate | 10 years
  Re-hospitalization of acute decompensated heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Dachun Xu, PhD, Principal Investigator — Shanghai Tenthth People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Su Y, Ma M, Zhang H, Pan X, Zhang X, Zhang F, Lv Y, Yan C. Prognostic value of serum hyponatremia for outcomes in patients with heart failure with preserved ejection fraction: An observational cohort study. Exp Ther Med. 2020 Nov;20(5):101. doi: 10.3892/etm.2020.9231. Epub 2020 Sep 17. PMID 32973950